CLINICAL TRIAL: NCT00338923
Title: Wound Healing Effects of HO/03/03 In Patients With Diabetic Neuropathic Plantar and Venous Ulcers, Pilot Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HealOr (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO-01-05
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Diabetic Foot Ulcer; Venous Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

ARMS (1):
- Treatment arm (Active Comparator): One Arm - Active Compound (HO/03/03)
  Interventions: Drug: HO/03/03

INTERVENTIONS:
Drug: HO/03/03

SUMMARY:
This is a multicenter pilot study to assess the healing effects of HO/03/03 on diabetic neuropathic plantar and venous ulcers.

HO/03/03 action mechanism involves the manipulation of keratinocyte and fibroblast migration and differentiation at the wound area.

* The primary end point of this study is assessment of safety in treating with HO/03/03 and the efficacy of the drug to promote wound closure of chronic wounds.
* The secondary end points are assessment time to closure and healing rate for the measurement of wound healing progression.

DETAILED DESCRIPTION:
This is a multicenter pilot study to assess the healing effects of HO/03/03 on diabetic neuropathic plantar and venous ulcers.

Pretreatment phase: During a pretreatment phase that will last up to 14 days, all patients will receive the conventional treatment once a day at the discretion of the investigator. All wounds will be morphologically monitored by photo documentation daily and measurements of wound area once a week.

Initial study visit: patients will begin treatment after completing all necessary demands in pre-treatment phase or after ruling out of all exclusion criteria. All wounds will be cleaned from previous treatment by surgical debridement and irrigation (saline).

Treatment phase: Following the pre-treatment phase, wounds will be treated topically with HO/03/03 for 30 days. During this 30 day phase, patients will receive daily treatments with HO/03/03 either at home by a certified nurse or at the clinic. Wounds will be monitored by certified medical staff member as well as photo documentation. Then application of the treatment followed by a 15-minute rest. Finally wound will be dressed with a fresh dressing and monitoring of any adverse events.

Patients will be administered HO/03/03 in addition to weight off-load Once a week wounds will be monitored by a physician: wounds size will be determined and documented. Patients will be evaluated for pain sensation at the wound area by filling a pain scoring questionnaire.

Twice during the experiment patients will undergo blood profile, HbA1c, blood glucose, and urine samples testing at the initial and terminating visits.

At the conclusion of the treatment phase the following will be completed:

* A physical examination;
* Collection of all blood and urine samples for clinical laboratory tests (dip sticks);

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following inclusion criteria to be included in the study:

1. be male or female over the age of 18;
2. have a diabetic neuropathic plantar and/or venous ulcer;
3. wound diameter <10cm;
4. wound depth is no more than exposed muscle;
5. have a current physical examination, which reveals no clinically significant abnormalities, except diabetes or diabetic ulcer/wound related condition
6. be available for the entire study period, and be able and willing to adhere to protocol requirements;
7. vascular inflow as measured by Doppler: ABI >= 0.7
8. have a debilitating wound over a period of 1 month prior to the experiment;
9. if female of childbearing potential, must be using a reliable form of birth control;
10. provide written informed consent prior to admission into the study.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following exclusion criteria:

1. have a body mass index (BMI) > 45;
2. have a glycosylated hemoglobin (HbAlc) > 12.0%;
3. have a history or presence of HIV or a clinically significant cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease;
4. have any clinically significant illness during the 4 weeks prior to admission into the study, except diabetes type1 or type2;
5. patients on concomitant medications that alter blood glucose levels (e.g., ACE inhibitors, lipid lowering agents, etc) must be on a stable dosage regimen for at least 4 weeks prior to entry into the study and the dosage must remain stable throughout the study;
6. patients on chemotherapy;
7. participation in a clinical study or use of an investigational drug within 30 days prior to admission to this study;
8. are pregnant or lactating;
9. visible bone exposure at wound site;
10. have any signs of clinical infection in the wound (which could be linked to raised body temperature), necrosis, erythema or mild drainage;
11. have any acute illness within 2 weeks prior to Screening;
12. residing in a nursing facility and/or are bed-ridden (unable to come to receive treatment at the clinic);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety | Treatment Period

SECONDARY OUTCOMES:
Time to Heal & Rate of Healing | Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: Micha Rapoport, Dr., Principal Investigator — Assaf Harofe Medical Center; Leon Gilead, Dr., Principal Investigator — Hadassah Ein Kerem Medical Center; Zvi Landau, Dr., Principal Investigator — Kaplan Medical Center
Locations (3):
- Israel (3):
  - Assaf Harofe Medical Center, Beer Yaakov
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot